CLINICAL TRIAL: NCT07327359
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Phase 1b/2a Study to Evaluate the Safety and Efficacy of OLX72021 in Healthy Males With Androgenetic Alopecia
Brief Title: A Study to Evaluate Safety and Efficacy of OLX72021 in Healthy Males With Androgenetic Alopecia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Olix Pharmaceuticals, Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLX72021-02
Record Dates: First submitted 2025-12-04; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: Male Pattern Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): Phase 1b : 2 dose level cohorts. Participants receive a total of 3 intradermal treatments of OLX72021 or placebo 28 days apart
  Interventions: Drug: OLX72021
- Phase 2a (Experimental): Phase 2a: 4 groups (1 group placebo and 3 groups with OLX72021). Participants receive 6 treatments of either placebo or OLX72021 via intradermal injection 28 days apart
  Interventions: Drug: OLX72021; Drug: Placebo

INTERVENTIONS:
Drug: OLX72021 — Low Dose
  Arms: Phase 2a
Drug: OLX72021 — Mid Dose
Drug: OLX72021 — High Dose
Drug: Placebo — Placebo
  Arms: Phase 2a

SUMMARY:
This study is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of OLX72021 in medically healthy men with mild to moderate androgenetic alopecia.

DETAILED DESCRIPTION:
This is a Phase 1b/2a double-blind, randomized, placebo-controlled, multiple ascending dose study evaluating the safety, efficacy, and pharmacokinetics (PK) of OLX72021 at a maximum of 2 dose levels. In Phase 1b, evaluation of dose levels will be conducted in a sequential manner with lower dose levels evaluated first in the sequence. Each dose level will be evaluated in a cohort of 12 participants with 9 participants receiving OLX72021 and 3 participants receiving placebo, approximately 24 participants in total. Cohorts may be dosed concurrently in Phase 2a. Each dose level will be evaluated in approximately 134 participants receiving OLX72021 or placebo for Phase 2a.

ELIGIBILITY:
Inclusion Criteria:

* Adult male.
* 18 to 59 years.
* Androgenetic Alopecia (Hamilton-Norwood III-V).
* Body mass index (BMI) ≥ 18.0 kg/m2, with a body weight ≥ 50 kg at screening.
* Non-smoker.
* Medically healthy without clinically significant abnormalities.
* Willing and able to tolerate multiple injections and attend all study visits.
* Willing to have blood drawn.

Exclusion Criteria:

* History or presence of significant pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant.
* Uncontrolled diabetes mellitus.
* Immunodeficiency disorders.
* History of clinically significant heart disease.
* History of risk factors for torsade de pointes.
* Any dermatological disorders of the scalp.
* History or clinical signs of keloids or hypertrophic scars.
* History of active hair loss due to alopecia areata, scarring alopecia, diffuse telogen effluvium, or conditions other than AGA.
* History of surgical correction of hair loss or hair transplant on the scalp.
* History of radiation of the scalp at any time.
* Use of semi-permanent hair products.
* Use of an occlusive wig, hair extensions, or hair weaves for the duration of the study.
* Use of cosmeceuticals or over-the-counter (OTC) hair regrowth products < 2 weeks prior to the first dose of study drug.
* Use of topical/local treatments.
* Use of non-topical/local medications within 24 weeks prior to the first dose of study drug
* Anti-cancer agents, including cytotoxic agents, that can potentially have effects on alopecia within 12 months prior to the first dose of study drug
* Scalp hair loss on the treatment area due to disease, injury, or medical therapy.
* Current infection that requires systemically absorbed or topical antibiotic, antifungal, antiparasitic, or antiviral medications.
* Any history of malignant disease in the last 5 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
* Positive test results for active human immunodeficiency virus-1 or 2 (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies.
* Positive drugs of abuse test, alcohol breath test, or cotinine test at the screening visit and prior to the first administration of study treatment.
* Use of any vaccinations within 14 days prior to the first study drug administration.
* Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.
* Treatment with an investigational drug in another clinical trial within 60 days or 5 half lives of the other investigational drug (whichever is longer) prior to the first administration of study drug in this trial.
* Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
* Known hypersensitivity to the study drug or any of the study drug ingredients.
* History of surgery or hospitalization within 3 months prior to screening, or surgery planned during the study.
* Regular consumption of more than 10 standard alcoholic drinks/week and/or more than 2 standard alcoholic drinks on any one day.
* Refusal to provide informed consent.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To investigate the incidence, type, severity, and relationship of adverse events (AEs)/serious AEs (SAEs), assessed using the CTCAE Version 5.0 (Phase 1b) | From baseline to end of study (Day 85)
To assess local tolerability at intradermal (ID) injection site (Phase 1b) | From baseline to end of study (Day 85)
To evaluate the change from baseline in non-vellus Target Area Hair Count (TAHC) at 24 weeks (Day 169) (Phase 2a) | Baseline to Day 169

SECONDARY OUTCOMES:
To measure time to plasma Cmax (Tmax) (Phase 1b) | From baseline to Day 58
To measure maximum observed plasma concentration (Cmax) (Phase 1b) | From baseline to Day 58
To measure area under the plasma concentration-time curve from 0 to time of last quantifiable concentration (AUClast) (Phase 1b) | From baseline to Day 58
To measure area under the plasma concentration-time curve from 0 to infinity (AUCinf) (Phase 1b) | From baseline to Day 58
To measure apparent terminal elimination half-life (t1/2) (Phase 1b) | From baseline to Day 58
To measure total apparent body clearance (CL/F) (Phase 1b) | From baseline to Day 58
To measure apparent volume of distribution (Vz/F) (Phase 1b) | From baseline to Day 58
To evaluate the change from baseline in non-vellus Target Area Hair Count (TAHC) at Day 29, Day 57, Day 85, Day 113, and Day 141 (Phase 2a) | From baseline to Day 141
To investigate the incidence, type, severity, and relationship of adverse events (AEs)/serious AEs (SAEs) (Phase 2a) | From baseline to end of study (Day 169)
To investigate the local tolerability at intradermal (ID) injection site (Phase 2a) | From baseline to end of study (Day 169)

CONTACTS AND LOCATIONS:
Locations (1):
- Emeritus Research Camberwell, Camberwell, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No